CLINICAL TRIAL: NCT00134719
Title: A Multicentre Primary & Booster Vaccination Study of GSK Biologicals' Hib-MenCY-TT Conjugate Vaccine vs ActHIB® & MenC Conjugate Licensed Vaccine When Given According to the 2-4-6 Month Schedule to Healthy Infants With Booster Dose at 12 to 15 Months
Brief Title: Hib-MenCY-TT Vaccine Study Compared to Licensed Hib and Meningococcal Serogroup C Conjugate Vaccines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 102370 (primary study); 102371 (Other: GSK); NCT00787046 (obsolete NCT alias)
Record Dates: First submitted 2005-08-10; First posted 2005-08-25 (Estimated); Results first posted 2012-07-20 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-05

CONDITIONS: Neisseria Meningitidis; Haemophilus Influenzae Type b
Keywords: Invasive Hib & N. meningitidis diseases
MeSH Terms: conditions — Haemophilus Infections | interventions — Hib-MenCY-TT vaccine; Heptavalent Pneumococcal Conjugate Vaccine; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate; Chickenpox Vaccine; Haemophilus influenzae-type b polysaccharide-Neisseria meningitidis outer membrane protein conjugate vaccine

ARMS (3):
- MenHibrix Group (Experimental): Subjects primed in study 102370 with 3 doses of MenHibrix, Infanrix Penta and Prevenar vaccines and receiving a fourth dose of MenHibrix co-administered with M-M-RII and Varivax vaccines in study 102371.
  Interventions: Biological: MenHibrix (Hib-MenCY-TT); Biological: Infanrix® Penta; Biological: Prevenar®; Biological: M-M-R®II; Biological: Varivax®
- ActHIB + Meningitec Group (Active Comparator): Subjects primed in study 102370 with 3 doses of ActHIB, Infanrix Penta, Prevenar and Meningitec vaccines and receiving a dose of MenHibrix co-administered with M-M-RII and Varivax vaccines in study 102371.
  Interventions: Biological: MenHibrix (Hib-MenCY-TT); Biological: Infanrix® Penta; Biological: Prevenar®; Biological: ActHIB®; Biological: Meningitec®; Biological: M-M-R®II; Biological: Varivax®
- ActHIB/PedvaxHIB Group (Active Comparator): Subjects primed in study 102370 with 3 doses of ActHIB, Infanrix Penta and Prevenar vaccines and receiving a dose of PedvaxHIB co-administered with M-M-RII and Varivax vaccines in study 102371.
  Interventions: Biological: Infanrix® Penta; Biological: Prevenar®; Biological: ActHIB®; Biological: M-M-R®II; Biological: Varivax®; Biological: PedvaxHIB®

INTERVENTIONS:
Biological: MenHibrix (Hib-MenCY-TT) — One intramuscular dose at 2, 4 and 6 months of age ( group A) and one intramuscular dose at 12 to 15 months of age (groups A and B)
  Arms: ActHIB + Meningitec Group; MenHibrix Group
Biological: Infanrix® Penta — One intramuscular dose at 2, 4 and 6 months of age
Biological: Prevenar® — One intramuscular dose at 2, 4 and 6 months of age
Biological: ActHIB® — One intramuscular dose at 2, 4 and 6 months of age
  Arms: ActHIB + Meningitec Group; ActHIB/PedvaxHIB Group
Biological: Meningitec® — One intramuscular dose at 2, 4 and 6 months of age
  Arms: ActHIB + Meningitec Group
Biological: M-M-R®II — One subcutaneous dose at 12-15 months of age
Biological: Varivax® — One subcutaneous dose at 12 to 15 months of age
Biological: PedvaxHIB® — One intramuscular dose at 12 to 15 months of age
  Arms: ActHIB/PedvaxHIB Group

SUMMARY:
This study is evaluating the safety and immunogenicity of Hib-MenCY-TT vaccine compared to control groups receiving licensed Hib or MenC conjugate vaccines, each administered at 2, 4, 6, and 12 to 15 months of age. Co-administration with live, attenuated measles, mumps, and rubella combination vaccine; and with live, attenuated varicella vaccine will be assessed with administration of the booster dose. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, September 2007.

DETAILED DESCRIPTION:
The study will be conducted in 2 stages: a 3-dose primary vaccination at 2, 4 and 6 months of age and a booster vaccination at 12 to 15 months of age. All subjects will have 3 blood samples taken. Half of the subjects of each group will have a blood sample taken just prior to the administration of the third dose of the primary vaccination and the other half of the subjects of each group will have a blood sample taken at one month after the third vaccine dose of the primary vaccination phase. In addition, all subjects of all groups will have a blood sample taken before and 42 days after administration of the booster dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Born after a gestation period between 36 and 42 weeks.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine(s).
* Previous vaccination against Neisseria meningitidis, Haemophilus influenzae type b, diphtheria, tetanus, pertussis, poliovirus, and/or Streptococcus pneumoniae; more than one previous dose of hepatitis B vaccine. Vaccination with hepatitis B at birth is accepted (although not mandatory). Influenza vaccination is allowed 30 days after administration of the third vaccine dose to 30 days preceding the booster dose.
* History of Neisseria meningitidis, Haemophilus influenzae type b, diphtheria, tetanus, pertussis, hepatitis B, poliovirus, Streptococcus pneumoniae and/or varicella invasive disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s), including dry natural latex rubber, tetanus toxoid, diphtheria toxoid, neomycin, polymyxin.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Additional specific criteria for the booster part of the study
* History of or previous vaccination against measles, mumps, rubella or varicella.
* Previous booster vaccination with Hib or meningococcal serogroup C vaccine since the last visit of the primary phase.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1104 (Actual)
Dates: Start 2005-04-11 (Actual); Primary Completion 2006-07-24 (Actual); Study Completion 2007-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Australia (3):
  - GSK Investigational Site, North Adelaide, South Australia
  - GSK Investigational Site, Carlton, Victoria
  - GSK Investigational Site, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bryant KA, Marshall GS. Haemophilus influenzae type b-Neisseria meningitidis serogroups C and Y tetanus toxoid conjugate vaccine for infants and toddlers. Expert Rev Vaccines. 2011 Jul;10(7):941-50. doi: 10.1586/erv.11.90. PMID 21806393
- [Background] Bryant K, McVernon J, Marchant C, Nolan T, Marshall G, Richmond P, Marshall H, Nissen M, Lambert S, Aris E, Mesaros N, Miller J. Immunogenicity and safety of measles-mumps-rubella and varicella vaccines coadministered with a fourth dose of Haemophilus influenzae type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine in toddlers: a pooled analysis of randomized trials. Hum Vaccin Immunother. 2012 Aug;8(8):1036-41. doi: 10.4161/hv.20357. Epub 2012 Aug 1. PMID 22617844
- [Background] Nolan T, Richmond P, Marshall H, McVernon J, Alexander K, Mesaros N, Aris E, Miller J, Poolman J, Boutriau D. Immunogenicity and safety of an investigational combined haemophilus influenzae type B-Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine. Pediatr Infect Dis J. 2011 Mar;30(3):190-6. doi: 10.1097/INF.0b013e3181fcb2bf. PMID 20948453
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 102370 (primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 102370 (primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 102370 (primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 102370 (primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 102370 are summarised with study 102371 on the GSK Clinical Study Register.
- Available data/document: Study Protocol: 102370 (primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomised at the beginning of the primary vaccination phase and kept their group assignment during the fourth dose vaccination phase. Not all subjects who completed the primary vaccination phase returned for participation in the fourth dose vaccination phase.
Pre-assignment Details: One subject who had a subject number allocated, was not vaccinated.
Period: Primary Vaccination Phase
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Started | 661 | 221 | 221
Completed | 647 | 215 | 216
Not Completed | 14 | 6 | 5
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 2
Not completed — Lost to Follow-up | 7 | 3 | 3
Period: Fourth Dose Vaccination Phase
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Started | 625 | 206 | 204
Completed | 623 | 203 | 203
Not Completed | 2 | 3 | 1
Not completed — Lost to Follow-up | 1 | 3 | 1
Not completed — Mother just delivered a new baby | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group | Total
Number analyzed (Participants) | 661 | 221 | 221 | 1103
Age, Continuous [Mean (Standard Deviation); unit: Days] | 61.0 (7.38) | 61.5 (7.22) | 61.5 (7.95) | 61.2 (7.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 328 | 118 | 103 | 549
  Male | 333 | 103 | 118 | 554

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-polyribosyl-ribitol-phosphate (Anti-PRP) Concentration Greater Than or Equal to 1.0 Microgram Per Milliliter (µg/mL)
Description: The analysis was performed on blood samples taken from half of the subjects in the MenHibrix and ActHIB/PedvaxHib groups only. The other half of the subjects in these study groups donated a blood sample after the second vaccine dose for analysis of the corresponding secondary outcome measure.
Time Frame: One month after the 3-dose primary vaccination course
Population: Analysis was performed on half of the subjects in the MenHibrix and ActHIB/PedvaxHib groups only, on the Primary According-to-Protocol (ATP) Cohort for Immunogenicity, including all evaluable subjects with assay result available for the considered time point.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 265 | 0 | 90
Participants | 255 |  | 76

2. Primary Outcome: Number of Subjects With Meningococcal Polysaccharide C Serum Bactericidal Activity/Assay Using Baby Rabbit Complement (rSBA-MenC) Titer Greater Than or Equal to 1:128
Description: The analysis was performed on blood samples taken from half of the subjects in the MenHibrix and ActHIB + Meningitec groups only. The other half of the subjects in these study groups donated a blood sample after the second vaccine dose for analysis of the corresponding secondary outcome measure.
Time Frame: One month after the 3-dose primary vaccination course
Population: Analysis was performed on subjects in the MenHibrix and ActHIB + Meningitec groups only, on the Primary According-to-Protocol Cohort for Immunogenicity, including all evaluable subjects with assay result available for the considered time point.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 287 | 99 | 0
Participants | 271 | 95 |

3. Primary Outcome: Number of Subjects Seroconverted for Anti-measles Antibodies
Description: The analysis was performed on blood samples taken from the subjects in the MenHibrix and ActHIB groups only. Anti-measles seroconversion is defined as the appearance of antibodies (i.e. concentration greater than or equal to the cut-off value of 150 milli-international units per milliliter (mIU/mL)) in the serum of subjects seronegative (below 150 mIU/mL) before vaccination.
Time Frame: 42 days after the fourth dose vaccination
Population: Analysis was performed on initially seronegative subjects in the MenHibrix and ActHIB groups only, on the Fourth dose According-to-Protocol cohort for immunogenicity, including all evaluable subjects with assay result available for the blood sample taken at 42 days after the administration of the fourth vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 852 | 0 | 286
Participants | 815 |  | 274

4. Primary Outcome: Number of Subjects Seroconverted for Anti-mumps Antibodies
Description: The analysis was performed on blood samples taken from the subjects in the MenHibrix and ActHIB groups only. Anti-mumps seroconversion is defined as titer greater than or equal to 28 ED50 in subjects seronegative (<28 ED50) before vaccination.
  ED50 is defined as the reciprocal of the sample dilution in the neutralising assay reducing the number of viral plaques by fifty percent.
Time Frame: 42 days after the fourth dose vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 601 | 0 | 191
Participants | 595 |  | 191

5. Primary Outcome: Number of Subjects With an Anti-rubella Seroresponse
Description: The analysis was performed on blood samples taken from the subjects in the MenHibrix and ActHIB groups only. Anti-rubella seroresponse is defined as post-vaccination concentration greater than or equal to 10 IU/mL (ELISA, Enzygnost) in subjects seronegative (concentration below 4 IU/mL) before vaccination.
Time Frame: 42 days after the fourth dose vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 850 | 0 | 285
Participants | 848 |  | 284

6. Primary Outcome: Number of Subjects Seroconverted for Anti-varicella Antibodies
Description: The analysis was performed on blood samples taken from the subjects in the MenHibrix and ActHIB groups only. Anti-varicella seroconversion is defined as post-vaccination titers greater than or equal to 1:5, in subjects seronegative (titers below 1:5) before vaccination.
Time Frame: 42 days after the fourth dose vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 723 | 0 | 223
Participants | 722 |  | 223

7. Secondary Outcome: Number of Subjects With rSBA-MenC Titer Greater Than or Equal to Pre-defined Cut-off Values
Description: The analyses for post-Dose 2 and post-Dose 3 data were performed on blood samples taken from the respective half of the subjects at both time points. The cut-off values assessed were titers 1:8 and 1:128.
Time Frame: After the second vaccine dose (post-dose 2), one month after the 3-dose primary vaccination course (post-dose 3), just prior to (pre-dose 4) and 42 days after the fourth dose (post-dose 4)
Population: Analysis was performed on the Primary ATP Cohort for Immunogenicity (post-Dose 2 and post-Dose 3), the ATP Cohort for Persistence (pre-Dose 4) and the Fourth Dose ATP Cohort for Immunogenicity (post-Dose 4), including all evaluable subjects with assay result available for the considered time point.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 496 | 169 | 164
Participants
  Post-dose 2 titer ≥ 1:8: number analyzed (Participants) | 295 | 100 | 92
  Post-dose 2 titer ≥ 1:8 | 282 | 97 | 2
  Post-dose 3 titer ≥ 1:8: number analyzed (Participants) | 287 | 99 | 99
  Post-dose 3 titer ≥ 1:8 | 284 | 99 | 5
  Pre-dose 4 titer ≥ 1:8: number analyzed (Participants) | 495 | 169 | 164
  Pre-dose 4 titer ≥ 1:8 | 449 | 143 | 16
  Post-dose 4 titer ≥ 1:8: number analyzed (Participants) | 496 | 162 | 157
  Post-dose 4 titer ≥ 1:8 | 494 | 155 | 16
  Post-dose 2 titer ≥ 1:128: number analyzed (Participants) | 295 | 100 | 92
  Post-dose 2 titer ≥ 1:128 | 239 | 91 | 0
  Post-dose 3 titer ≥ 1:128: number analyzed (Participants) | 287 | 99 | 99
  Post-dose 3 titer ≥ 1:128 | 271 | 95 | 0
  Pre-dose 4 titer ≥ 1:128: number analyzed (Participants) | 495 | 169 | 164
  Pre-dose 4 titer ≥ 1:128 | 241 | 50 | 1
  Post-dose 4 titer ≥ 1:128: number analyzed (Participants) | 496 | 162 | 157
  Post-dose 4 titer ≥ 1:128 | 482 | 115 | 5

8. Secondary Outcome: rSBA-MenC Titers
Description: The analyses for post-Dose 2 and post-Dose 3 data were performed on blood samples taken from the respective half of the subjects at both time points. Titers are given as Geometric Mean Titers.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 496 | 169 | 164
titer
  Post-dose 2: number analyzed (Participants) | 295 | 100 | 92
  Post-dose 2 | 356.9 [302.6 to 420.9] | 714.5 [541.6 to 942.7] | 4.2 [3.9 to 4.5]
  Post-dose 3: number analyzed (Participants) | 287 | 99 | 99
  Post-dose 3 | 804.6 [699.9 to 924.9] | 790.1 [649.4 to 961.2] | 4.5 [4.0 to 5.0]
  Pre-dose 4: number analyzed (Participants) | 495 | 169 | 164
  Pre-dose 4 | 102.8 [90.1 to 117.3] | 53.7 [43.0 to 67.1] | 5.2 [4.6 to 5.9]
  Post-dose 4: number analyzed (Participants) | 496 | 162 | 157
  Post-dose 4 | 1696.7 [1515.8 to 1899.2] | 261.9 [204.4 to 335.7] | 5.4 [4.7 to 6.2]

9. Secondary Outcome: Number of Subjects With rSBA-MenY Titer Greater Than or Equal to Pre-defined Cut-off Values
Description: as for outcome 7
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 514 | 167 | 159
Participants
  Post-dose 2 titer ≥ 1:8: number analyzed (Participants) | 293 | 99 | 92
  Post-dose 2 titer ≥ 1:8 | 289 | 10 | 13
  Post-dose 3 titer ≥ 1:8: number analyzed (Participants) | 288 | 98 | 97
  Post-dose 3 titer ≥ 1:8 | 287 | 16 | 22
  Pre-dose 4 titer ≥ 1:8 | 506 | 65 | 42
  Post-dose 4 titer ≥ 1:8: number analyzed (Participants) | 496 | 164 | 157
  Post-dose 4 titer ≥ 1:8 | 496 | 162 | 90
  Post-dose 2 titer ≥ 1:128: number analyzed (Participants) | 293 | 99 | 92
  Post-dose 2 titer ≥ 1:128 | 224 | 2 | 3
  Post-dose 3 titer ≥ 1:128: number analyzed (Participants) | 288 | 98 | 97
  Post-dose 3 titer ≥ 1:128 | 264 | 9 | 5
  Pre-dose 4 titer ≥ 1:128 | 414 | 35 | 19
  Post-dose 4 titer ≥ 1:128: number analyzed (Participants) | 496 | 164 | 157
  Post-dose 4 titer ≥ 1:128 | 493 | 152 | 59

10. Secondary Outcome: rSBA-MenY Titers
Description: as for outcome 8
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 514 | 167 | 159
Titer
  Post-dose 2: number analyzed (Participants) | 293 | 99 | 92
  Post-dose 2 | 315.6 [271.6 to 366.9] | 5.4 [4.5 to 6.5] | 5.9 [4.7 to 7.3]
  Post-dose 3: number analyzed (Participants) | 288 | 98 | 97
  Post-dose 3 | 728.3 [635.5 to 834.7] | 7.1 [5.4 to 9.3] | 7.7 [5.9 to 10.2]
  Pre-dose 4 | 264.4 [240.7 to 290.4] | 16.0 [12.0 to 21.2] | 10.5 [8.0 to 13.6]
  Post-dose 4: number analyzed (Participants) | 496 | 164 | 157
  Post-dose 4 | 1986.5 [1825.9 to 2161.3] | 797.7 [658.5 to 966.2] | 34.4 [25.2 to 47.0]

11. Secondary Outcome: Number of Subjects With Meningococcal Polysaccharide C Serum Bactericidal Activity/Assay Using Human Complement (hSBA-MenC) Antibody Titer Greater Than or Equal to Pre-defined Cut-off Values
Description: The analysis for was performed on the first 30% of the blood samples taken at each time point. The cut-off values assessed were titers 1:4 and 1:8.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 134 | 54 | 50
Participants
  Post-dose 2 titer ≥ 1:4: number analyzed (Participants) | 89 | 31 | 25
  Post-dose 2 titer ≥ 1:4 | 85 | 29 | 0
  Post-dose 3 titer ≥ 1:4: number analyzed (Participants) | 83 | 28 | 28
  Post-dose 3 titer ≥ 1:4 | 83 | 28 | 0
  Pre-dose 4 titer ≥ 1:4 | 125 | 46 | 5
  Post-dose 4 titer ≥ 1:4: number analyzed (Participants) | 132 | 43 | 46
  Post-dose 4 titer ≥ 1:4 | 131 | 41 | 1
  Post-dose 2 titer ≥ 1:8: number analyzed (Participants) | 89 | 31 | 25
  Post-dose 2 titer ≥ 1:8 | 84 | 29 | 0
  Post-dose 3 titer ≥ 1:8: number analyzed (Participants) | 83 | 28 | 28
  Post-dose 3 titer ≥ 1:8 | 83 | 28 | 0
  Pre-dose 4 titer ≥ 1:8 | 125 | 46 | 5
  Post-dose 4 titer ≥ 1:8: number analyzed (Participants) | 132 | 43 | 46
  Post-dose 4 titer ≥ 1:8 | 131 | 41 | 1

12. Secondary Outcome: hSBA-MenC Titers
Description: The analysis for was performed on the first 30% of the blood samples taken at each time point. Titers are given as Geometric Mean Titers.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 134 | 54 | 50
Titer
  Post-dose 2: number analyzed (Participants) | 89 | 31 | 25
  Post-dose 2 | 179.4 [130.3 to 247.1] | 319.0 [173.6 to 586.2] | 2.0 [2.0 to 2.0]
  Post-dose 3: number analyzed (Participants) | 83 | 28 | 28
  Post-dose 3 | 379.4 [294.6 to 488.6] | 254.2 [192.7 to 335.4] | 2.0 [2.0 to 2.0]
  Pre-dose 4 | 97.7 [74.0 to 128.9] | 34.6 [22.8 to 52.6] | 2.6 [2.0 to 3.3]
  Post-dose 4: number analyzed (Participants) | 132 | 43 | 46
  Post-dose 4 | 1807.6 [1398.2 to 2336.8] | 171.5 [94.7 to 310.8] | 2.2 [1.8 to 2.6]

13. Secondary Outcome: Number of Subjects With Meningococcal Polysaccharide Y Serum Bactericidal Activity/Assay Using Human Complement (hSBA-MenY) Antibody Titer Greater Than or Equal to Pre-defined Cut-off Values
Description: as for outcome 11
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 122 | 44 | 41
Participants
  Post-dose 2 titer ≥ 1:4: number analyzed (Participants) | 88 | 31 | 25
  Post-dose 2 titer ≥ 1:4 | 79 | 0 | 0
  Post-dose 3 titer ≥ 1:4: number analyzed (Participants) | 85 | 28 | 29
  Post-dose 3 titer ≥ 1:4 | 85 | 0 | 0
  Pre-dose 4 titer ≥ 1:4: number analyzed (Participants) | 114 | 44 | 41
  Pre-dose 4 titer ≥ 1:4 | 104 | 1 | 0
  Post-dose 4 titer ≥ 1:4: number analyzed (Participants) | 122 | 34 | 35
  Post-dose 4 titer ≥ 1:4 | 119 | 15 | 16
  Post-dose 2 titer ≥ 1:8: number analyzed (Participants) | 88 | 31 | 25
  Post-dose 2 titer ≥ 1:8 | 73 | 0 | 0
  Post-dose 3 titer ≥ 1:8: number analyzed (Participants) | 85 | 28 | 29
  Post-dose 3 titer ≥ 1:8 | 85 | 0 | 0
  Pre-dose 4 titer ≥ 1:8: number analyzed (Participants) | 114 | 44 | 41
  Pre-dose 4 titer ≥ 1:8 | 103 | 1 | 0
  Post-dose 4 titer ≥ 1:8: number analyzed (Participants) | 122 | 34 | 35
  Post-dose 4 titer ≥ 1:8 | 119 | 13 | 16

14. Secondary Outcome: hSBA-MenY Titers
Description: as for outcome 12
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 122 | 44 | 41
Titer
  Post-dose 2: number analyzed (Participants) | 88 | 31 | 25
  Post-dose 2 | 25.6 [19.3 to 34.1] | 2.0 [2.0 to 2.0] | 2.0 [2.0 to 2.0]
  Post-dose 3: number analyzed (Participants) | 85 | 28 | 29
  Post-dose 3 | 86.4 [68.9 to 108.3] | 2.0 [2.0 to 2.0] | 2.0 [2.0 to 2.0]
  Pre-dose 4: number analyzed (Participants) | 114 | 44 | 41
  Pre-dose 4 | 81.2 [58.6 to 112.6] | 2.2 [1.8 to 2.7] | 2.0 [2.0 to 2.0]
  Post-dose 4: number analyzed (Participants) | 122 | 34 | 35
  Post-dose 4 | 1002.2 [740.9 to 1355.7] | 8.8 [4.4 to 17.3] | 18.3 [7.7 to 43.6]

15. Secondary Outcome: Number of Subjects With Anti-Polysaccharide C (Anti-PSC) Antibody Concentration Greater Than or Equal to Pre-defined Cut-off Values
Description: The analysis for post-Dose 2 and post-Dose 3 data was performed on blood samples taken from the respective half of the subjects at both time points. The cut-off values assessed were 0.3 µg/mL and 2 µg/mL.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 490 | 160 | 138
Participants
  Post-dose 2 concentration ≥0.3 µg/mL: number analyzed (Participants) | 296 | 95 | 85
  Post-dose 2 concentration ≥0.3 µg/mL | 296 | 95 | 7
  Post-dose 3 concentration ≥0.3 µg/mL: number analyzed (Participants) | 276 | 95 | 91
  Post-dose 3 concentration ≥0.3 µg/mL | 276 | 95 | 3
  Pre-dose 4 concentration≥0.3 µg/mL: number analyzed (Participants) | 475 | 160 | 138
  Pre-dose 4 concentration≥0.3 µg/mL | 417 | 138 | 2
  Post-dose 4 concentration≥0.3µg/mL: number analyzed (Participants) | 490 | 160 | 122
  Post-dose 4 concentration≥0.3µg/mL | 489 | 158 | 1
  Post-dose 2 concentration ≥2.0 µg/mL: number analyzed (Participants) | 296 | 95 | 85
  Post-dose 2 concentration ≥2.0 µg/mL | 248 | 81 | 1
  Post-dose 3 concentration ≥2.0 µg/mL: number analyzed (Participants) | 276 | 95 | 91
  Post-dose 3 concentration ≥2.0 µg/mL | 241 | 79 | 0
  Pre-dose 4 concentration≥2.0 µg/mL: number analyzed (Participants) | 475 | 160 | 138
  Pre-dose 4 concentration≥2.0 µg/mL | 53 | 31 | 0
  Post-dose 4 concentration≥2.0µg/mL: number analyzed (Participants) | 490 | 160 | 122
  Post-dose 4 concentration≥2.0µg/mL | 408 | 95 | 0

16. Secondary Outcome: Anti-PSC Concentrations
Description: The analysis for post-Dose 2 and post-Dose 3 data was performed on blood samples taken from the respective half of the subjects at both time points. Concentrations are given as Geometric Mean Concentrations.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter (µg/mL)
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 490 | 160 | 138
Microgram per milliliter (µg/mL)
  Post-dose 2: number analyzed (Participants) | 296 | 95 | 85
  Post-dose 2 | 4.32 [3.98 to 4.69] | 3.54 [3.08 to 4.06] | 0.17 [0.15 to 0.19]
  Post-dose 3: number analyzed (Participants) | 276 | 95 | 91
  Post-dose 3 | 4.15 [3.87 to 4.46] | 3.94 [3.40 to 4.55] | 0.16 [0.15 to 0.17]
  Pre-dose 4: number analyzed (Participants) | 475 | 160 | 138
  Pre-dose 4 | 0.77 [0.71 to 0.83] | 0.86 [0.73 to 1.01] | 0.15 [0.15 to 0.16]
  Post-dose 4: number analyzed (Participants) | 490 | 160 | 122
  Post-dose 4 | 4.78 [4.42 to 5.16] | 2.65 [2.24 to 3.14] | 0.15 [0.15 to 0.16]

17. Secondary Outcome: Number of Subjects With Anti-Polysaccharide Y (Anti-PSY) Antibody Concentration Greater Than or Equal to Pre-defined Cut-off Values
Description: as for outcome 15
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 502 | 162 | 122
Participants
  Post-dose 2 concentration ≥0.3 µg/mL: number analyzed (Participants) | 291 | 92 | 83
  Post-dose 2 concentration ≥0.3 µg/mL | 291 | 3 | 6
  Post-dose 3 concentration ≥0.3 µg/mL: number analyzed (Participants) | 269 | 91 | 88
  Post-dose 3 concentration ≥0.3 µg/mL | 269 | 3 | 4
  Pre-dose 4 concentration≥0.3 µg/mL: number analyzed (Participants) | 474 | 136 | 112
  Pre-dose 4 concentration≥0.3 µg/mL | 469 | 2 | 4
  Post-dose 4 concentration≥0.3µg/mL | 502 | 160 | 3
  Post-dose 2 concentration ≥2.0 µg/mL: number analyzed (Participants) | 291 | 92 | 83
  Post-dose 2 concentration ≥2.0 µg/mL | 268 | 0 | 0
  Post-dose 3 concentration ≥2.0 µg/mL: number analyzed (Participants) | 269 | 91 | 88
  Post-dose 3 concentration ≥2.0 µg/mL | 266 | 0 | 0
  Pre-dose 4 concentration≥2.0 µg/mL: number analyzed (Participants) | 474 | 136 | 112
  Pre-dose 4 concentration≥2.0 µg/mL | 278 | 1 | 2
  Post-dose 4 concentration≥2.0µg/mL | 96 | 46 | 1

18. Secondary Outcome: Anti-PSY Concentrations
Description: as for outcome 16
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter (µg/mL)
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 502 | 162 | 122
Microgram per milliliter (µg/mL)
  Post-dose 2: number analyzed (Participants) | 291 | 92 | 83
  Post-dose 2 | 7.81 [7.04 to 8.67] | 0.16 [0.15 to 0.16] | 0.17 [0.15 to 0.19]
  Post-dose 3: number analyzed (Participants) | 269 | 91 | 88
  Post-dose 3 | 12.92 [11.80 to 14.14] | 0.15 [0.15 to 0.16] | 0.16 [0.15 to 0.17]
  Pre-dose 4: number analyzed (Participants) | 474 | 136 | 112
  Pre-dose 4 | 2.44 [2.26 to 2.64] | 0.16 [0.15 to 0.16] | 0.16 [0.15 to 0.18]
  Post-dose 4 | 16.92 [15.60 to 18.35] | 7.09 [6.05 to 8.31] | 0.16 [0.15 to 0.17]

19. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentration Greater Than or Equal to Pre-defined Cut-off Values
Description: The analysis for post-Dose 2 and post-Dose 3 data was performed on blood samples taken from the respective half of the subjects at both time points. The cut-off values assessed were 0.15 µg/mL and 1.0 µg/mL.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 562 | 189 | 182
Participants
  Post-dose 2 ≥ 0.15 µg/mL: number analyzed (Participants) | 280 | 94 | 85
  Post-dose 2 ≥ 0.15 µg/mL | 255 | 77 | 70
  Post-dose 3 ≥ 0.15 µg/mL: number analyzed (Participants) | 265 | 88 | 90
  Post-dose 3 ≥ 0.15 µg/mL | 265 | 85 | 88
  Pre-dose 4 ≥ 0.15 µg/mL: number analyzed (Participants) | 562 | 189 | 181
  Pre-dose 4 ≥ 0.15 µg/mL | 541 | 160 | 159
  Post-dose 4 ≥ 0.15 µg/mL: number analyzed (Participants) | 549 | 185 | 182
  Post-dose 4 ≥ 0.15 µg/mL | 549 | 183 | 182
  Post-dose 2 ≥ 1.0 µg/mL: number analyzed (Participants) | 280 | 94 | 85
  Post-dose 2 ≥ 1.0 µg/mL | 151 | 41 | 40
  Post-dose 3 ≥ 1.0 µg/mL: number analyzed (Participants) | 265 | 88 | 90
  Post-dose 3 ≥ 1.0 µg/mL | 255 | 74 | 76
  Pre-dose 4 ≥ 1.0 µg/mL: number analyzed (Participants) | 562 | 189 | 181
  Pre-dose 4 ≥ 1.0 µg/mL | 314 | 71 | 74
  Post-dose 4 ≥ 1.0 µg/mL: number analyzed (Participants) | 549 | 185 | 182
  Post-dose 4 ≥ 1.0 µg/mL | 547 | 176 | 179

20. Secondary Outcome: Anti-PRP Concentrations
Description: as for outcome 16
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter (µg/mL)
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 562 | 189 | 182
Microgram per milliliter (µg/mL)
  Post-dose 2: number analyzed (Participants) | 280 | 94 | 85
  Post-dose 2 | 1.320 [1.097 to 1.588] | 0.788 [0.571 to 1.089] | 0.861 [0.607 to 1.222]
  Post-dose 3: number analyzed (Participants) | 265 | 88 | 90
  Post-dose 3 | 8.551 [7.502 to 9.746] | 3.692 [2.747 to 4.961] | 5.014 [3.675 to 6.841]
  Pre-dose 4: number analyzed (Participants) | 562 | 189 | 181
  Pre-dose 4 | 1.175 [1.061 to 1.300] | 0.668 [0.544 to 0.820] | 0.748 [0.611 to 0.916]
  Post-dose 4: number analyzed (Participants) | 549 | 185 | 182
  Post-dose 4 | 34.890 [31.687 to 38.417] | 13.442 [11.057 to 16.343] | 20.975 [17.668 to 24.899]

21. Secondary Outcome: Number of Subjects With Anti-measles Concentration Greater Than or Equal to 150 mIU/mL
Description: The cut-off value assessed was 150 mIU/mL.
Time Frame: Just prior to the fourth dose and 42 days after the fourth dose
Population: Analysis was performed on the Fourth Dose ATP Cohort for Immunogenicity, including all evaluable subjects with assay result available for the considered time point.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 542 | 185 | 178
Participants
  Just prior to the fourth dose: number analyzed (Participants) | 513 | 174 | 175
  Just prior to the fourth dose | 0 | 1 | 0
  42 days after the fourth dose | 510 | 173 | 170

22. Secondary Outcome: Number of Subjects With Anti-mumps Titer Greater Than or Equal to 24 ED50
Description: ED50 is defined as the reciprocal of the sample dilution in the neutralising assay reducing the number of viral plaques by fifty percent.
Time Frame: Just prior to the fourth dose and 42 days after the fourth dose
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 509 | 170 | 165
Participants
  Just prior to the fourth dose: number analyzed (Participants) | 494 | 165 | 159
  Just prior to the fourth dose | 179 | 59 | 52
  42 days after the fourth dose | 505 | 169 | 163

23. Secondary Outcome: Number of Subjects With Anti-rubella Concentration Greater Than or Equal to 4 IU/mL
Description: The cut-off value assessed was 4 IU/mL.
Time Frame: Just prior to the fourth dose and 42 days after the fourth dose
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 540 | 185 | 177
Participants
  Just prior to the fourth dose: number analyzed (Participants) | 516 | 175 | 176
  Just prior to the fourth dose | 2 | 1 | 0
  42 days after the fourth dose | 540 | 184 | 177

24. Secondary Outcome: Number of Subjects With Anti-varicella Titer Greater Than or Equal to 1:5
Description: The cut-off value assessed was a titer of 1:5.
Time Frame: Just prior to the fourth dose and 42 days after the fourth dose
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 548 | 184 | 179
Participants
  Just prior to the fourth dose: number analyzed (Participants) | 533 | 181 | 177
  Just prior to the fourth dose | 126 | 44 | 56
  42 days after the fourth dose | 547 | 183 | 179

25. Secondary Outcome: Number of Subjects With a Fourth Dose Response for hSBA-MenC
Description: Fourth dose response for hSBA-MenC is defined as: •For initially seronegative subjects (i.e., subjects with pre fourth dose hSBA antibody titer below 1:4), post fourth dose hSBA antibody titer greater than or equal to 1:16; •For initially seropositive subjects (i.e., subjects with pre fourth dose antibody titer greater than or equal to 1:4), post fourth dose hSBA antibody titer greater than or equal to 1:128.
Time Frame: 42 days after the fourth dose
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 103 | 36 | 40
Participants | 100 | 23 | 1

26. Secondary Outcome: Number of Subjects With a Fourth Dose Response for hSBA-MenY
Description: Fourth dose response for hSBA-MenY defined as: •For initially seronegative subjects (i.e., pre fourth dose hSBA antibody titer < 1:4), post fourth dose hSBA antibody titer greater than or equal to (≥) 1:16; •For initially seropositive subjects with pre fourth dose hSBA antibody titer ≥ 1:4 and < 1:64, post fourth dose hSBA antibody titer at least 4-fold higher than the pre fourth dose hSBA antibody titer; •For initially seropositive subjects with pre fourth dose hSBA antibody titer ≥ 1:64, post fourth dose hSBA antibody titer at least 2-fold higher than the pre fourth dose hSBA antibody titer.
Time Frame: 42 days after the fourth dose
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 81 | 23 | 29
Participants | 75 | 6 | 16

27. Secondary Outcome: Number of Subjects With Anti-measles Concentration Greater Than or Equal to Predefined Cut-off Values in Initially Seronegative Subjects
Description: The pre-defined cut-off values were 150 mIU/mL and 200 mIU/mL. Initially seronegative subjects are defined as subjects with pre-vaccination anti-measles concentration below 150 mIU/mL.
Time Frame: 42 days after the fourth dose
Population: Analysis was performed on initially seronegative subjects in the Fourth Dose ATP Cohort for Immunogenicity, including all evaluable subjects with assay result available for the considered time point.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 501 | 173 | 171
Participants
  Greater than or equal to 150 mIU/mL | 469 | 164 | 163
  Greater than or equal to 200 mIU/mL | 466 | 163 | 162

28. Secondary Outcome: Anti-measles Concentrations in Initially Seronegative Subjects
Description: Concentrations are presented as Geometric Mean Concentrations expressed as mIU/mL. Initially seronegative subjects are defined as subjects with pre-vaccination anti-measles concentration below 150 mIU/mL.
Time Frame: 42 days after the fourth dose
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Milli-International Units per Milliliter
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 501 | 173 | 171
Milli-International Units per Milliliter | 1627.494 [1469.996 to 1801.866] | 1773.293 [1500.779 to 2095.292] | 1786.404 [1523.083 to 2095.250]

29. Secondary Outcome: Number of Subjects With Anti-rubella Concentration Greater Than or Equal to Predefined Cut-off Values in Initially Seronegative Subjects
Description: The pre-defined cut-off values were 4 IU/mL and 10 IU/mL. Initially seronegative subjects are defined as subjects with pre-vaccination anti-measles concentration below 4 IU/mL.
Time Frame: 42 days after the fourth dose
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 500 | 174 | 171
Participants
  ≥ 4 International Units per Milliliter | 500 | 174 | 171
  ≥ 10 International Units per Milliliter | 498 | 173 | 171

30. Secondary Outcome: Anti-rubella Concentrations in Initially Seronegative Subjects
Description: Concentrations are presented as Geometric Mean Concentrations expressed as IU/mL. Initially seronegative subjects are defined as subjects with pre-vaccination anti-rubella concentration below 4 IU/mL.
Time Frame: 42 days after the fourth dose
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: International Units per Milliliter
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 500 | 174 | 171
International Units per Milliliter | 78.779 [73.941 to 83.932] | 83.168 [74.535 to 92.801] | 76.691 [69.019 to 85.217]

31. Secondary Outcome: Number of Subjects With Anti-mumps Titer Greater Than or Equal to 28 ED50 in Subjects With Anti-mumps Titer Below 28 ED50 Before Vaccination
Description: as for outcome 22
Time Frame: 42 days after the fourth dose
Population: Analysis was performed on subjects with a pre-vaccination anti-mumps titer below 28 ED50 in the Fourth Dose ATP Cohort for Immunogenicity, including all evaluable subjects with assay result available for the considered time point.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 332 | 115 | 110
Participants | 330 | 115 | 110

32. Secondary Outcome: Number of Subjects With Anti-mumps Titer Greater Than or Equal to Predefined Cut-off Values in Initially Seronegative Subjects
Description: The pre-defined cut-off values were 28 ED50 and 51 ED50. Initially seronegative subjects are defined as subjects with pre-vaccination anti-mumps titer below 24 ED50.
Time Frame: 42 days after the fourth dose
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 293 | 98 | 102
Participants
  Greater than or equal to 28 ED50 | 293 | 98 | 102
  Greater than or equal to 51 ED50 | 265 | 92 | 93

33. Secondary Outcome: Anti-mumps Titers in Initially Seronegative Subjects
Description: Titers are presented as Geometric Mean Titers expressed as ED50, the reciprocal of the sample dilution in the neutralising assay reducing the number of viral plaques by fifty percent. Initially seronegative subjects are defined as subjects with pre-vaccination anti-mumps titer below 24 ED50.
Time Frame: 42 days after the fourth dose
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 293 | 98 | 102
Titer | 120.777 [111.967 to 130.281] | 145.405 [128.318 to 164.766] | 115.279 [101.835 to 130.498]

34. Secondary Outcome: Number of Subjects With Anti-varicella Titer Greater Than or Equal to Predefined Cut-off Values in Initially Seronegative Subjects
Description: The pre-defined cut-off values were 1:5 and 1:40. Initially seronegative subjects are defined as subjects with pre-vaccination anti-varicella titer below 1:5.
Time Frame: 42 days after the fourth dose
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 404 | 136 | 119
Participants
  Titer greater than or equal to 1:5 | 403 | 136 | 119
  Titer greater than or equal to 1:40 | 403 | 136 | 119

35. Secondary Outcome: Anti-varicella Titers in Initially Seronegative Subjects
Description: Titers are presented as Geometric Mean Titers. Initially seronegative subjects are defined as subjects with pre-vaccination anti-varicella titer below 1:5.
Time Frame: 42 days after the fourth dose
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 404 | 136 | 119
Titer | 414.633 [391.361 to 439.288] | 468.985 [421.845 to 521.393] | 438.280 [394.261 to 487.214]

36. Secondary Outcome: Number of Subjects Reporting Solicited Local and General Symptoms During the Primary Vaccination Phase
Description: Solicited local symptoms assessed include pain, redness and swelling. Solicited general symptoms assessed include drowsiness, fever (rectal temperature greater than or equal to 38 degrees Celcius), irritability and loss of appetite.
Time Frame: During a 4-day period (Day 0-3) after any vaccine dose in the primary vaccination phase
Population: Analysis was performed on all subjects with an available symptom sheet in the Primary Total Vaccinated Cohort, including all subjects vaccinated during the primary vaccination phase.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 659 | 220 | 220
Participants
  Pain | 432 | 171 | 152
  Redness | 556 | 189 | 189
  Swelling | 492 | 163 | 167
  Drowsiness | 530 | 193 | 176
  Fever | 196 | 83 | 80
  Irritability | 616 | 211 | 212
  Loss of appetite | 410 | 153 | 135

37. Secondary Outcome: Number of Subjects Reporting Solicited Local and General Symptoms During the Fourth Dose Vaccination Phase
Description: as for outcome 36
Time Frame: During a 4-day period (Day 0-3) after the fourth dose vaccination phase
Population: Analysis was performed on all subjects with an available symptom sheet in the Fourth Dose Total Vaccinated Cohort, including all subjects vaccinated during the fourth dose vaccination phase.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 622 | 202 | 201
Participants
  Pain | 217 | 60 | 100
  Redness | 379 | 102 | 157
  Swelling | 225 | 63 | 123
  Drowsiness | 196 | 63 | 71
  Fever | 60 | 14 | 31
  Irritability | 361 | 120 | 117
  Loss of appetite | 224 | 76 | 62

38. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events
Description: Unsolicited adverse event covers any adverse event reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-day (Day 0-30) post-primary and post-fourth dose vaccination period
Population: Analysis was performed on the Primary Total Vaccinated Cohort and the Fourth Dose Total Vaccinated Cohort, including all subjects vaccinated during the primary and fourth dose vaccination phases, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 661 | 221 | 221
Participants
  Post-primary vaccination period | 490 | 166 | 158
  Post-fourth dose vaccination period | 429 | 139 | 147

39. Secondary Outcome: Number of Subjects Reporting Specific Solicited General AEs Related to Measles, Mumps, Rubella Vaccine and Varicella Vaccine
Description: Specific solicited general symptoms assessed include fever (temperature greater than or equal to 38 degrees Celcius), meningismus/ febrile convulsion, parotid / salivary gland swelling and rash.
Time Frame: During a 43-day (Day 0-42) after the fourth dose
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 622 | 202 | 201
Participants
  Fever | 324 | 107 | 112
  Meningismus/ febrile convulsion | 0 | 0 | 0
  Parotid / salivary gland swelling | 4 | 1 | 0
  Rash | 232 | 86 | 66

40. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs), New Onset of Chronic Illnesses (NOCI), Rash, Emergency Room Visits (ER), Physician Office Visits (PO) During the Primary Vaccination Phase
Description: SAEs: medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. NOCI: e.g. autoimmune disorders, asthma, type I diabetes and allergies. Types of rash: hives, idiopathic thrombocytopenic purpura and petechiae. ER and PO visits assessed were not related to well-child care, vaccination, injury or common acute illnesses such as upper respiratory tract infection, otitis media, pharyngitis and gastroenteritis.
Time Frame: From enrolment through the day preceding the fourth dose
Population: Analysis was performed on the Primary Total Vaccinated Cohort, including all subjects vaccinated during the primary vaccination phase.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 661 | 221 | 221
Participants
  Rash | 176 | 67 | 51
  New onset of chronic illnesses | 124 | 39 | 36
  Emergency room visits | 81 | 22 | 14
  Physician office visits | 291 | 90 | 88
  Serious adverse events | 55 | 21 | 15

41. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs), New Onset of Chronic Illnesses (NOCI), Rash, Emergency Room Visits (ER), Physician Office Visits (PO) During the Fourth Dose Vaccination Phase
Description: as for outcome 40
Time Frame: From the day of administration of the fourth dose until the end of the extended safety follow-up period (last study contact at 18-21 months of age
Population: Analysis was performed on the Fourth Dose Total Vaccinated Cohort, including all subjects vaccinated during the ourth dose vaccination phase.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Number analyzed (Participants) | 625 | 206 | 204
Participants
  Rash | 52 | 15 | 13
  New onset of chronic illnesses | 20 | 8 | 5
  Emergency room visits | 42 | 13 | 10
  Physician office visits | 220 | 64 | 63
  Serious adverse events | 40 | 12 | 8

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs): From Day 0 up to 18-21 months of age; Non-systematically assessed frequent AEs: Day 0-30 post-primary and post-fourth dose; Systematically assessed frequent AEs: Day 0-3 post-primary and post-fourth dose vaccination phase.
Description: SAEs and non-systematically assessed frequent AEs were assessed on the Primary & Fourth dose Total Vaccinated Cohort, respectively. Systematically assessed frequent AEs were assessed on respectively subjects from the Primary and Fourth dose Total Vaccinated Cohort who returned their symptom sheet.
Arm/Group | MenHibrix Group | ActHIB + Meningitec Group | ActHIB/PedvaxHIB Group
Serious Adverse Events (participants affected / at risk) | 55/661 | 21/221 | 15/221
Other Adverse Events (participants affected / at risk) | 657/661 | 220/221 | 220/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | MenHibrix Group (N=661) | ActHIB + Meningitec Group (N=221) | ActHIB/PedvaxHIB Group (N=221)
Cyanosis (Cardiac disorders) | 1 | 0 | 0 — Post-primary vaccination phase
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 — Post-primary vaccination phase
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 1 | 0 — Post-primary vaccination phase
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1 — Post-primary vaccination phase
Respiratory tract malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0 — Post-primary vaccination phase
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 — Post-primary vaccination phase
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 — Post-primary vaccination phase
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 — Post-primary vaccination phase
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 — Post-primary vaccination phase
Food allergy (Immune system disorders) | 1 | 0 | 1 — Post-primary vaccination phase
Bronchiolitis (Infections and infestations) | 6 | 3 | 5 — Post-primary vaccination phase
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0 — Post-primary vaccination phase
Croup infectious (Infections and infestations) | 3 | 1 | 0 — Post-primary vaccination phase
Escherichia urinary tract infection (Infections and infestations) | 2 | 0 | 0 — Post-primary vaccination phase
Exanthema subitum (Infections and infestations) | 1 | 0 | 0 — Post-primary vaccination phase
Gastroenteritis (Infections and infestations) | 9 | 3 | 2 — Post-primary vaccination phase
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 — Post-primary vaccination phase
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 — Post-primary vaccination phase
Otitis media (Infections and infestations) | 5 | 2 | 1 — Post-primary vaccination phase
Otitis media chronic (Infections and infestations) | 1 | 0 | 0 — Post-primary vaccination phase
Perianal abscess (Infections and infestations) | 1 | 0 | 0 — Post-primary vaccination phase
Pneumonia (Infections and infestations) | 2 | 1 | 1 — Post-primary vaccination phase
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0 — Post-primary vaccination phase
Pneumonia primary atypical (Infections and infestations) | 0 | 1 | 0 — Post-primary vaccination phase
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 — Post-primary vaccination phase
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 | 1 | 0 — Post-primary vaccination phase
Sepsis (Infections and infestations) | 1 | 1 | 0 — Post-primary vaccination phase
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 — Post-primary vaccination phase
Tonsillitis (Infections and infestations) | 0 | 1 | 0 — Post-primary vaccination phase
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 — Post-primary vaccination phase
Urinary tract infection (Infections and infestations) | 4 | 0 | 0 — Post-primary vaccination phase
Viral infection (Infections and infestations) | 1 | 3 | 1 — Post-primary vaccination phase
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 — Post-primary vaccination phase
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Post-primary vaccination phase
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 — Post-primary vaccination phase
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Post-primary vaccination phase
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 — Post-primary vaccination phase
Investigation (Investigations) | 0 | 0 | 1 — Post-primary vaccination phase
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0 — Post-primary vaccination phase
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Post-primary vaccination phase
Epilepsy (Nervous system disorders) | 1 | 0 | 0 — Post-primary vaccination phase
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0 — Post-primary vaccination phase
Hypotonic-hyporesponsive episode (Nervous system disorders) | 1 | 0 | 0 — Post-primary vaccination phase
Infantile spasms (Nervous system disorders) | 0 | 0 | 1 — Post-primary vaccination phase
Breath holding (Psychiatric disorders) | 1 | 0 | 0 — Post-primary vaccination phase
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0 | 0 — Post-primary vaccination phase
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 — Post-primary vaccination phase
Joint effusion (Musculoskeletal and connective tissue disorders) | 1/625 | 0/206 | 0/204 — Post-fourth dose vaccination phase
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/625 | 0/206 | 0/204 — Post-fourth dose vaccination phase
Febrile convulsion (Nervous system disorders) | 2/625 | 1/206 | 0/204 — Post-fourth dose vaccination phase
Asthma (Respiratory, thoracic and mediastinal disorders) | 4/625 | 1/206 | 0/204 — Post-fourth dose vaccination phase
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1/625 | 0/206 | 1/204 — Post-fourth dose vaccination phase
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3/625 | 1/206 | 0/204 — Post-fourth dose vaccination phase
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — Post-primary vaccination phase
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Post-primary vaccination phase
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Post-primary vaccination phase
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Post-primary vaccination phase
Supraventricular tachycardia (Cardiac disorders) | 0/625 | 0/206 | 1/204 — Post-fourth dose vaccination phase
Middle ear effusion (Ear and labyrinth disorders) | 1/625 | 0/206 | 0/204 — Post-fourth dose vaccination phase
Otorrhoea (Ear and labyrinth disorders) | 0/625 | 0/206 | 1/204 — Post-fourth dose vaccination phase
Oesophageal rupture (Gastrointestinal disorders) | 1/625 | 0/206 | 0/204 — Post-fourth dose vaccination phase
Bronchiolitis (Infections and infestations) | 1/625 | 0/206 | 2/204 — Post-fourth dose vaccination phase
Croup infectious (Infections and infestations) | 2/625 | 0/206 | 0/204 — Post-fourth dose vaccination phase
Gastroenteritis (Infections and infestations) | 11/625 | 0/206 | 1/204 — Post-fourth dose vaccination phase
Gastroenteritis rotavirus (Infections and infestations) | 3/625 | 0/206 | 0/204 — Post-fourth dose vaccination phase
Gastroenteritis viral (Infections and infestations) | 0/625 | 1/206 | 0/204 — Post-fourth dose vaccination phase
Otitis media (Infections and infestations) | 8/625 | 1/206 | 0/204 — Post-fourth dose vaccination phase
Otitis media chronic (Infections and infestations) | 0/625 | 1/206 | 0/204 — Post-fourth dose vaccination phase
Pharyngeal abscess (Infections and infestations) | 0/625 | 1/206 | 0/204 — Post-fourth dose vaccination phase
Pneumonia viral (Infections and infestations) | 1/625 | 1/206 | 0/204 — Post-fourth dose vaccination phase
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0/625 | 3/206 | 1/204 — Post-fourth dose vaccination phase
Tonsillitis (Infections and infestations) | 2/625 | 0/206 | 0/204 — Post-fourth dose vaccination phase
Upper respiratory tract infection (Infections and infestations) | 1/625 | 1/206 | 0/204 — Post-fourth dose vaccination phase
Urinary tract infection (Infections and infestations) | 0/625 | 0/206 | 1/204 — Post-fourth dose vaccination phase
Viral infection (Infections and infestations) | 1/625 | 0/206 | 0/204 — Post-fourth dose vaccination phase
Viral tonsillitis (Infections and infestations) | 1/625 | 0/206 | 0/204 — Post-fourth dose vaccination phase
Viral upper respiratory tract infection (Infections and infestations) | 1/625 | 0/206 | 0/204 — Post-fourth dose vaccination phase
Accidental exposure (Injury, poisoning and procedural complications) | 1/625 | 0/206 | 0/204 — Post-fourth dose vaccination phase
Drug toxicity (Injury, poisoning and procedural complications) | 1/625 | 0/206 | 0/204 — Post-fourth dose vaccination phase
Mouth injury (Injury, poisoning and procedural complications) | 1/625 | 0/206 | 0/204 — Post-fourth dose vaccination phase
Thermal burn (Infections and infestations) | 0/625 | 0/206 | 1/204 — Post-fourth dose vaccination phase
Tooth fracture (Injury, poisoning and procedural complications) | 0/625 | 1/206 | 0/204 — Post-fourth dose vaccination phase
Dehydration (Metabolism and nutrition disorders) | 1/625 | 0/206 | 0/204 — Post-fourth dose vaccination phase
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | MenHibrix Group (N=661) | ActHIB + Meningitec Group (N=221) | ActHIB/PedvaxHIB Group (N=221)
Pain at the injection site (General disorders) | 432/658 | 171/220 | 152/220 — This post-primary vaccination phase solicited local symptom was assessed in subjects who had symptom sheet filled in.
Redness at the injection site (General disorders) | 556/658 | 189/220 | 189/220 — This post-primary vaccination phase solicited local symptom was assessed in subjects who had symptom sheet filled in.
Swelling at the injection site (General disorders) | 492/658 | 163/220 | 167/220 — This post-primary vaccination phase solicited local symptom was assessed in subjects who had symptom sheet filled in.
Pain at the injection site (General disorders) | 217/622 | 60/202 | 100/201 — This post-fourth dose vaccination phase solicited local symptom was assessed in subjects who had symptom sheet filled in.
Redness at the injection site (General disorders) | 379/622 | 102/202 | 157/201 — This post-fourth dose vaccination phase solicited local symptom was assessed in subjects who had symptom sheet filled in.
Swelling at the injection site (General disorders) | 225/622 | 63/202 | 123/201 — This post-fourth dose vaccination phase solicited local symptom was assessed in subjects who had symptom sheet filled in.
Drowsiness (General disorders) | 530/659 | 193/220 | 176/220 — This post-primary vaccination phase solicited general symptom was assessed in subjects who had symptom sheet filled in.
Fever (General disorders) | 196/659 | 83/220 | 80/220 — This post-primary vaccination phase solicited general symptom was assessed in subjects who had symptom sheet filled in.
Irritability (General disorders) | 616/659 | 211/220 | 212/220 — This post-primary vaccination phase solicited general symptom was assessed in subjects who had symptom sheet filled in.
Loss of appetite (General disorders) | 410/659 | 153/220 | 135/220 — This post-primary vaccination phase solicited general symptom was assessed in subjects who had symptom sheet filled in.
Drowsiness (General disorders) | 196/622 | 63/202 | 71/201 — This post-fourth dose vaccination phase solicited general symptom was assessed in subjects who had symptom sheet filled in.
Fever (General disorders) | 60/622 | 14/202 | 31/201 — This post-fourth dose vaccination phase solicited general symptom was assessed in subjects who had symptom sheet filled in.
Irritability (General disorders) | 361/622 | 120/202 | 117/201 — This post-fourth dose vaccination phase solicited general symptom was assessed in subjects who had symptom sheet filled in.
Loss of appetite (General disorders) | 224/622 | 76/202 | 62/201 — This post-fourth dose vaccination phase solicited general symptom was assessed in subjects who had symptom sheet filled in.
Upper respiratory tract infection (Infections and infestations) | 154 | 53 | 54 — Post-primary vaccination phase
Injection site bruising (General disorders) | 98 | 44 | 27 — Post-primary vaccination phase
Teething (Gastrointestinal disorders) | 99 | 33 | 26 — Post-primary vaccination phase
Vomiting (Gastrointestinal disorders) | 52 | 16 | 15 — Post-primary vaccination phase
Eczema (Skin and subcutaneous tissue disorders) | 49 | 16 | 17 — Post-primary vaccination phase
Rash (Skin and subcutaneous tissue disorders) | 49 | 20 | 10 — Post-primary vaccination phase
Irritability (General disorders) | 48 | 12 | 14 — Post-primary vaccination phase
Injection site nodule (General disorders) | 44 | 14 | 10 — Post-primary vaccination phase
Pyrexia (General disorders) | 37 | 9 | 18 — Post-primary vaccination phase
Diarrhea (Gastrointestinal disorders) | 40 | 10 | 8 — Post-primary vaccination phase
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 24 | 4 | 17 — Post-primary vaccination phase
Upper respiratory tract infection (Infections and infestations) | 157/625 | 40/206 | 49/204 — Post-fourth dose vaccination phase
Teething (Gastrointestinal disorders) | 109/625 | 41/206 | 38/204 — Post-fourth dose vaccination phase
Irritability (General disorders) | 78/625 | 35/206 | 23/204 — Post-fourth dose vaccination phase
Diarrhoea (Gastrointestinal disorders) | 55/625 | 17/206 | 16/204 — Post-fourth dose vaccination phase
Otitis media (Infections and infestations) | 51/625 | 14/206 | 14/204 — Post-fourth dose vaccination phase
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 44/625 | 20/206 | 17/204 — Post-fourth dose vaccination phase
Vomiting (Gastrointestinal disorders) | 48/625 | 16/206 | 16/204 — Post-fourth dose vaccination phase
Injection site bruising (General disorders) | 41/625 | 14/206 | 17/204 — Post-fourth dose vaccination phase
Cough (Respiratory, thoracic and mediastinal disorders) | 24/625 | 9/206 | 13/204 — Post-fourth dose vaccination phase

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.